CLINICAL TRIAL: NCT03586258
Title: Anatomical Clinical Correlations. Neuropsychological and Brain Medical Imaging Study in Brain Damage Subjects 2 (CORAC2)
Brief Title: Neuropsychological and Brain Medical Imaging Study in Patients With Brain Damage 2
Acronym: CORAC2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-A03062-51; 2017-A03062-51 (Other: ANSM)
Record Dates: First submitted 2018-07-03; First posted 2018-07-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-01

CONDITIONS: Cerebrovascular Disorders; Brain Lesion; Degenerative Disease; Developmental Disability
Keywords: Neuropsychological study; Brain imaging
MeSH Terms: conditions — Cerebrovascular Disorders; Developmental Disabilities | interventions — Neuropsychological Tests; Neuroimaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brain Damaged Subjects (Experimental): Patients with circumscribed brain injury, developmental pathology or degenerative pathology responsible for selective cognitive disorders
  Interventions: Behavioral: Neuropsychological testing; Other: Brain Imaging; Other: Galvanic Vestibular Stimulation (GVS)
- Healthy Volunteers (Sham Comparator): Healthy Controls
  Interventions: Behavioral: Neuropsychological testing; Other: Brain Imaging; Other: Galvanic Vestibular Stimulation (GVS)

INTERVENTIONS:
Behavioral: Neuropsychological testing — Experimental test about cognitive deficit of interest and standard neuropsychological tests
Other: Brain Imaging — Anatomical, diffusion, and/or functional MRI
Other: Galvanic Vestibular Stimulation (GVS) — Stimulation versus Sham

SUMMARY:
Two groups of subjects will be constitute: (i) patients with circumscribed brain injury (including stroke, vascular malformations, tumor or circumscribed infectious lesions) or degenerative/developmental disorders and selective cognitive disorders; (ii) healthy control subjects.

The objective of this project is to evaluate specific neuropsychological deficits and apply current brain imaging techniques (anatomical, diffusion, functional, magnetic stimulation) to patients suffering from these cognitive deficits due to brain damage, in order to elucidate the brain mechanisms underlying these deficits.

ELIGIBILITY:
Inclusion Criteria:

* Age > 17 years
* French language
* Effective contraception for women during the study
* Informed consent
* No alcohol intake the day before the exam
* For patients only, focal cerebral lesion (stroke, malformation, tumor, inflammatory, infectious, traumatic), neonatal pathology, developmental or degenerative disease with cognitive deficit

Exclusion Criteria:

* For healthy volunteers: previous neurological history (except non complicated migraine or epilepsy), previous psychiatric history (except depression with good evolution or anxiety), or severe cranial traumatism
* For patients: vigilance disorders, severe depression or anxiety.
* For both: psychotropic medication other than a hypnotic or an anxiolytic at low doses without dose modification for at least one month, severe visual or auditory impairment, patient without judicial or administrative liberty, measure of legal protection or no capable to express their consent, pregnancy or breastfeeding, contraindication for MRI or GVS if applicable, participation in another trial or former involvement in another trial within one month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2019-01-10 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Cognitive Deficit | 3 months to more than 2 years
  The cognitive deficit of interest will depend on the localization of the brain lesion. The outcome measure could be a standardized neuropsychological test or an experimental test specifically elaborated for this protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier MARTINAUD, MD, PhD, Principal Investigator — Caen University Hospital, Normandie UNIV, UNICAEN, PSL Research University, EPHE, Inserm, U1077, CHU de Caen, Neuropsychologie et Imagerie de la Mémoire Humaine, 14000 Caen, France
Locations (1):
- Caen University Hospital, Caen, France